CLINICAL TRIAL: NCT03083431
Title: Oral Propranolol for Prevention of Threshold Retinopathy of Prematurity
Acronym: RoProp
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Ankara University (Other); University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RoProp; 32ER30_173677 (Other Grant/Funding Number: Swiss National Science Foundation (SNSF)); 2017-002124-24 (EudraCT Number)
Record Dates: First submitted 2017-03-13; First posted 2017-03-20 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind Placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propranolol (Experimental): Oral propranolol (1.6 mg propranolol-HCl/kg/d in 3-4 divided dosages) given for a maximum of 10 weeks (depending on postmenstrual gestational age at birth)
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator): Placebo (same duration as oral propranolol solution)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Oral propranolol (1.6 mg propranolol-hydrochloride/kg/d in 4 divided dosages)
  Arms: Propranolol
Drug: Placebo — Oral solution containing the same excipients as propranolol solution
  Arms: Placebo

SUMMARY:
Extremely premature infants are at risk of developing a potentially blinding eye disease, called retinopathy of prematurity (ROP). Currently available treatment, consisting of laser surgery or injection of drugs into the eye balls, may prevent most but not all cases of permanent ROP-mediated blindness. Both types of treatment are associated with significant costs and side effects.

An orally administered drug commonly used to treat hypertension, propranolol, may be effective in halting progression of ROP to severe stages, as suggested by preliminary data from small studies. As severe (threshold) ROP is an overall rare disease, the effectiveness of propranolol in combating ROP can only be assessed in a large, multicenter randomized controlled trial involving hospitals caring for extremely preterm infants of diverse origin.

DETAILED DESCRIPTION:
Threshold Retinopathy of Prematurity (ROP), observed in a fraction of extremely premature infants, is characterized by retinal vessel proliferation that threatens vision secondary to retinal detachment. Currently available treatments (ablative laser surgery or intravitreal anti-VEGF injections) may prevent most but not all cases of permanent ROP-mediated blindness and are associated with significant costs and side effects.

Orally administered propranolol, a commonly used drug to treat hypertension, may be effective in halting progression of ROP to severe stages, as suggested by preliminary data from small studies. Propranolol has been used for decades not only in adult patients but also in newborn infants with heart diseases. Moreover, it has been licensed in 2014 for the use in newborn infants with hemangioma in the European Union, Switzerland and the United States. This multicenter randomized placebo-controlled trial aims to assess whether oral propranolol given to extremely premature infants below 28 weeks gestational age reduces the rates of threshold ROP.

ELIGIBILITY:
Inclusion criteria:

* Preterm infant born before 28 week's gestation
* Birth weight below 1250 g
* At least 5 weeks of age (at randomisation)
* PMA 310/7 - 36 6/7 weeks
* Ophthalmoscopic evidence of incipient ROP (stage 1 or 2, with or without plus disease in any zone)
* Written informed consent by parents or legal guardian, according to national requirements

Exclusion Criteria:

* ROP stage ≥ 3, AP-ROP or suspected AP-ROP, or any other ROP requiring an intervention (study endpoint already reached).
* Conditions that indicate open label propranolol such as: thyrotoxicosis, arterial hypertension or certain heart diseases (such as tetralogy of Fallot, paroxysmal supraventricular tachycardia, or long QT syndrome) etc.
* Major congenital malformations or known chromosomal anomalies
* Colobomas and other eye malformations
* PHACE syndrome (posterior fossa anomalies, large infantile hemangiomas of the face, neck, and/or scalp, arterial lesions, cardiac abnormalities/coarctation of the aorta, eye anomalies) (risk of cerebrovascular complications)
* Very large hemangioma (risk of hyperkalemia), as judged by the attending physician
* Medication of the infant with rifampicin or phenobarbitone (enhanced metabolic clearance)
* Chronic kidney impairment (serum creatinine > 1.3 mg/dl [115 μmol/L])
* Severe liver dysfunction (ALT (GPT) > 900 U/L)
* Known hypersensitivity to propranolol or any of the excipients (see 6.3.1.)
* Prinzmetal's angina, Raynaud's phenomenon (severe peripheral arterial circulatory disturbance), or pheochromocytoma (contraindications for propranolol in adults, not occurring in newborn infants)
* Any circumstances that make the investigator believe that participation in the study leads to exceptional medical or organizational problems for the patient
* Conditions that prohibit propranolol therapy such as: Atrio-ventricular block grade 2 or 3 hypertrophic cardiomyopathy, sinoatrial block, uncontrolled heart failure or cardiogenic shock, bronchial asthma
* Medication of the infant or the mother if breastfeeding with clonidine, reserpine, angiotensin-converting enzyme inhibitors, angiotensin-receptor antagonists (contraindicated in preterm infants) or antiarrhythmic drugs including amiodarone, propafenone, lidocaine, digoxin/digitoxin, quinidine, verapamil, diltiazem, bepridil (pharmacodynamic interaction)

Ages: 5 Weeks to 15 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 276 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Survival without adverse ophthalmological outcome (stage ≥ 3, AP-ROP, or any ROP treatment) | 48 weeks postmenstrual age
  The primary endpoint for efficacy is survival until 48 weeks postmenstrual age without adverse ophthalmological outcome (stage ≥ 3, AP-ROP, or any ROP treatment) diagnosed according to the International Committee for the Classification of Retinopathy of Prematurity Revisited.

SECONDARY OUTCOMES:
Time to adverse ophthalmological outcome in days | 48 weeks postmenstrual age
  Time to adverse ophthalmological outcome in days (alternative to primary endpoint to account for the timing, considering death as a competing risk)
Survival without adverse ophthalmological outcome | 48 weeks postmenstrual age
  Survival without adverse ophthalmological outcome (as defined for the primary outcome)
Survival with adverse ophthalmological outcome | 48 weeks postmenstrual age
  Survival with adverse ophthalmological outcome (as defined for the primary outcome)
Survival without local treatment for ROP | 48 weeks postmenstrual age
  Survival without local treatment for ROP (ablative laser surgery or intravitreal injections of anti-VEGF agents).
Death until discharge | 48 weeks postmenstrual age
  Death until discharge
Death until 48 weeks postmenstrual age | 48 weeks postmenstrual age
  Death until 48 weeks postmenstrual age
Recurrence of ROP in infants treated with anti-VEGF-antagonists | 70 (+/- 2 weeks) postmenstrual age
  Recurrence of ROP in infants treated with anti-VEGF-antagonists
Need for repeated ROP therapy in infants treated with anti-VEGF-antagonists | 70 (+/- 2 weeks) postmenstrual age
  Need for repeated ROP therapy in infants treated with anti-VEGF-antagonists

OTHER OUTCOMES:
Intraventricular haemorrhages (all grades) | 48 weeks postmenstrual age
  Intraventricular haemorrhage (all grades)
Posthaemorrhagic hydrocephalus requiring intervention | 48 weeks postmenstrual age
  Posthaemorrhagic hydrocephalus requiring intervention
Cystic leukomalacia | 48 weeks postmenstrual age
  Cystic leukomalacia
Persistent ductus arteriosus requiring treatment | 48 weeks postmenstrual age
  Persistent ductus arteriosus requiring treatment
Bronchopulmonary dysplasia | 48 weeks postmenstrual age
  Bronchopulmonary dysplasia (mild, moderate, severe), defined and graded according to the consensus statement of the national institutes of health
Duration of subsequent hospitalisation | 48 weeks postmenstrual age
  Number of days of subsequent hospitalisations
Duration of primary hospitalisation | 48 weeks postmenstrual age
  Number of days of primary hospitalisation
Z-scores for weight | 48 weeks postmenstrual age
  Z-scores for weight at the beginning and end of IMP administration
Z-scores for head circumference | 48 weeks postmenstrual age
  Z-scores for head circumference at the beginning and end of IMP administration
Duration of supplemental oxygen | 48 weeks postmenstrual age
  Number of days on supplemental oxygen
Necrotizing enterocolitis | 48 weeks postmenstrual age
  Necrotizing enterocolitis (requiring surgery)
Safety: Culture-proven sepsis or meningitis during IMP administration | 48 weeks postmenstrual age
  Culture-proven sepsis or meningitis during IMP administration (defined as growth of a recognized pathogen not counting coagulase-negative staphylococci in blood or cerebrospinal fluid in an infant treated for at least 5 d with intravenous antibiotics and a rise of C-reactive protein to more than 10 mg/l during the first 72 h of antibiotic treatment)
Safety: Symptomatic hypoglycemia during IMP administration | 48 weeks postmenstrual age
  Symptomatic hypoglycemia during IMP administration (blood glucose < 30 mg/dl requiring intravenous glucose administration for 48 h or more), not counting glucose administration "to keep-vein-open" (e.g. at rates of ≤ 1 mL/h)
Safety: Emergency endotracheal intubation during IMP administration | 48 weeks postmenstrual age
  Emergency endotracheal intubation attributable to obstructive airway disease during IMP administration (excluding elective intubation for surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Bassler, M.D., Principal Investigator — University of Zurich
Locations (3):
- University Hospital Tübingen, Tübingen, Baden-Wurttemberg, Germany
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland
- Ankara University School of Medicine Children's Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data set containing gestational age (only weeks), birth weight (in 100g categories), year of birth, country, gender, intervention (propranolol or placebo), outcome (retinopathy of prematurity, maximum stage), date and type of treatment for retinopathy if any
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months - 5 years after publication of the results in a peer-reviewed journal
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee (learned intermediary)

REFERENCES:
- [Background] Buhrer C, Bassler D. Oral Propranolol: A New Treatment for Infants with Retinopathy of Prematurity? Neonatology. 2015;108(1):49-52. doi: 10.1159/000381659. Epub 2015 May 9. PMID 25968340
- [Background] Buhrer C, Erdeve O, Bassler D, Bar-Oz B. Oral propranolol for prevention of threshold retinopathy of prematurity (ROPROP): protocol of a randomised controlled trial. BMJ Open. 2018 Jul 6;8(7):e021749. doi: 10.1136/bmjopen-2018-021749. PMID 29982217